CLINICAL TRIAL: NCT05594251
Title: Early Detection of Endotheliopathy Post-Transplant
Status: Terminated | Type: Observational
Why Stopped: IRB approval 1/6/2025 to close to accrual with present enrollment. Project completed.
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Le Bonheur Children's Hospital (Other); University of Tennessee (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: EDEPT
Record Dates: First submitted 2022-10-14; First posted 2022-10-26 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Endotheliopathy
Keywords: Endotheliopathy; Early Detection; Post-Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this research study is to learn more about possible risk factors that might be associated with side effects from stem cell transplants in people between the ages of 0 to 26 years old. Specifically, this study is looking at complications that arise from injury to the endothelium, a small layer of cells lining the blood vessels and heart. These complications can affect the heart, lungs, liver, kidneys and intestines and increase risk of severe illness needing care in the intensive care unit.

DETAILED DESCRIPTION:
Primary Objectives:

* To evaluate the proportion of pediatric patients undergoing Hematopoietic cell transplantation (HCT) who develop critical illness (defined by admission to the pediatric intensive care unit at St. Jude for reasons other than observation after procedure) within 100 days of such therapies.
* To evaluate the proportion of pediatric patients undergoing HCT who experience development of endothelial-related organ dysfunction syndromes.

Secondary Objectives

* To report the baseline (pre-conditioning and post-conditioning but pre-cellular therapy) levels of specified circulating biomarkers, vascular reactivity as measured by reactive hyperemia index (RHI), and to describe baseline clot structure in patients age 0-26 years of age planned to undergo HCT.
* To compare the levels of circulating biomarkers between the cohort of patients that experience critical illness (defined by admission to the pediatric intensive care unit at St. Jude for reasons other than observation after procedure) any time during the first 100 days of HCT following cellular infusion and the cohort of patients that do not ever experience critical illness in the first 100 days of HCT following cellular infusion.
* To evaluate the time to development of any complications including development of endotheliopathies, development of critical illness (defined by admission to the pediatric intensive care unit at St. Jude for reasons other than observation after procedure), development of abnormal vascular reactivity by RHI, development of abnormal clot structure, and time to peak (or trough, if applicable) level of circulating biomarkers.

The study will require a minimum of 1 blood draw before transplant and 6 blood draws throughout the first 100 days following transplant. If participants are admitted to the intensive care unit or are diagnosed with specific complications additional blood draws will be done. Peripheral arterial tonometry (PAT) testing will occur 1-2 times during the first 100 days in several older patients who can tolerate the procedure by sitting still for the duration of the testing period.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-26 years planned to undergo allogeneic or autologous HCT for any indication with any preparative regimen planned.

Exclusion Criteria:

* Less than 10 kg at time of consent or any child in which blood volume required for scheduled blood draws would pose more than minimal risk.
* Lack of agreement from primary HCT physician.
* Inability or unwillingness of research participant and/or legal guardian/representative to give written informed consent.

Max Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants who meet the Eligibility Criteria
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Proportion of pediatric patients undergoing Hematopoietic cell transplantation (HCT) who develop critical illness | Up to 100 days after transplant (plus or minus 3 days)
  The proportion of pediatric patients undergoing HCT who develop critical illness (defined by admission to the pediatric intensive care unit at St. Jude for reasons other than observation after procedure) will be estimated using one-sample binomial estimates and various confidence intervals.
Proportion of pediatric patients undergoing HCT who experience development of endothelial-related organ dysfunction syndromes | Up to 100 days after transplant (plus or minus 3 days)
  The proportion will be estimated using one-sample binomial estimates and various confidence intervals.

SECONDARY OUTCOMES:
Baseline levels of circulating biomarkers | Baseline (before preparative transplant regimen starts) and Day 0 (on day of transplant, before therapy takes place)
  Descriptive statistics (mean, median, standard deviation) will be used.
Baseline vascular reactivity | Baseline (before preparative transplant regimen starts) and Day 0 (on day of transplant, before therapy takes place)
  Descriptive statistics (mean, median, standard deviation) will be used.
Baseline clot structure | Baseline (before preparative transplant regimen starts) and Day 0 (on day of transplant, before therapy takes place)
  Descriptive statistics (mean, median, standard deviation) will be used.
Difference in circulating biomarkers | From Baseline blood draws up to 100 days post ICU admission
  We will compare the levels of circulating biomarkers of patients that experience critical illness (defined by admission to the pediatric intensive care unit at St. Jude for reasons other than observation after procedure) and the patients that do not ever experience critical illness by using the linear mixed-effect model (LMM). Blood draws will be done at baseline, Day 0, and after transplant: days 1, 7, 14, 21, 28, 100 (plus or minus 3 days). Those with Endotheliopathy diagnosis anytime during the 100 days of HCT following cellular transfusion, and are admitted to ICU, will have additional blood draws: At the time of Endotheliopathy diagnosis (plus or minus 3 days), at the time of ICU admission (plus or minus 3 days), 72 hours after ICU admission (plus or minus 3 days), and every 7 days if remains admitted to the intensive care unit for longer than 72 hours (plus or minus 3 days) up to 100 days post ICU submission.
Difference in clot structure | From Baseline blood draws up to 100 days post ICU admission
  We will compare the clot structure of patients that experience critical illness (defined by admission to the pediatric intensive care unit at St. Jude for reasons other than observation after procedure) and the patients that do not ever experience critical illness by using the linear mixed-effect model (LMM). Blood draws will be done at baseline, Day 0, and after transplant: days 1, 7, 14, 21, 28, 100 (plus or minus 3 days). Those with Endotheliopathy diagnosis anytime during the 100 days of HCT following cellular transfusion, and are admitted to ICU, will have additional blood draws: At the time of Endotheliopathy diagnosis (plus or minus 3 days), at the time of ICU admission (plus or minus 3 days), 72 hours after ICU admission (plus or minus 3 days), and every 7 days if remains admitted to the intensive care unit for longer than 72 hours (plus or minus 3 days) up to 100 days post ICU submission.
Difference in vascular reactivity | From Baseline blood draws up to 100 days post ICU admission
  We will compare the vascular reactivity of patients that experience critical illness (defined by admission to the pediatric intensive care unit at St. Jude for reasons other than observation after procedure) and the patients that do not ever experience critical illness by using the linear mixed-effect model (LMM). Blood draws will be done at baseline, Day 0, and after transplant: days 1, 7, 14, 21, 28, 100 (plus or minus 3 days). Those with Endotheliopathy diagnosis anytime during the 100 days of HCT following cellular transfusion, and are admitted to ICU, will have additional blood draws: At the time of Endotheliopathy diagnosis (plus or minus 3 days), at the time of ICU admission (plus or minus 3 days), 72 hours after ICU admission (plus or minus 3 days), and every 7 days if remains admitted to the intensive care unit for longer than 72 hours (plus or minus 3 days) up to 100 days post ICU submission.
Time to development of any complications or critical illness | Up to 100 days after transplant (plus or minus 3 days)
  Will be assessed by the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Saad Ghafoor, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols